CLINICAL TRIAL: NCT03419091
Title: Prospective Trial of a Reusable Digital Flexible Ureteroscope vs a Single-Use Flexible Ureteroscope in the Treatment of Urolithiasis: An EDGE Consortium Clinical Trial
Brief Title: LithoVue Single Use Disposable Ureteroscope
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Ben Chew, MD, Associate Professor of Urology, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H16-02436
Record Dates: First submitted 2018-01-08; First posted 2018-02-01 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Kidney Stone
Keywords: ureteroscopy; lithovue; nephrolithiasis; single use ureteroscope
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis

STUDY DESIGN:
Intervention Model Description: This will be a prospective, randomized clinical trial. Patients will be randomized 1:1 in randomization blocks of 4 to undergo the procedure with either the LithoVue single use flexible ureteroscope or the digital reusable flexible ureteroscope. Ureteroscopy will be performed using a standardized technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Reusable Ureteroscope (Active Comparator): Standard ureteroscope.
  Interventions: Device: Reusable Ureteroscope
- single-use flexible digital ureteroscope (LithoVue) (Experimental): Disposable ureteroscope being tested.
  Interventions: Device: single-use flexible digital ureteroscope

INTERVENTIONS:
Device: single-use flexible digital ureteroscope — Device being tested.
  Other Names: LithoVue
  Arms: single-use flexible digital ureteroscope (LithoVue)
Device: Reusable Ureteroscope — Comparative device.
  Arms: Reusable Ureteroscope

SUMMARY:
Most flexible ureteroscopes that are used to treat kidney stones have been reusable. Recently, advances in technology have resulted in single-use (disposable) ureteroscopes to become available. The investigators are interested in determining if the performance of the two types of scopes are equivalent. This will help guide institutions in the future to purchase the best scopes for their patients.

DETAILED DESCRIPTION:
Ureteroscopy is commonly used in the treatment of kidney stones. Flexible ureteroscopes are costly to purchase and repair. Issues with flexible ureteroscopes include loss of deflection and visual performance (fiberoptic pixels) with use and the high repair costs. Reprocessing and sterilization of reusable ureteroscopes also requires staff who are specially trained and dedicated in this area. Inadequate sterilization could also lead to transmissible infections between patients. A single-use flexible digital ureteroscope has recently become commercially available (LithoVue, Boston Scientific, Marlborough, MA). Pre-clinical testing show the accessibility to the ureter and all areas of the kidney to be equivalent to current flexible ureteroscopes. However, clinical data comparing this single-use ureteroscope to a current state of the art reusable ureteroscope is lacking. Establishing at least equivalence in performance between the new single use ureteroscope and a reusable digital ureteroscope will help surgeons and operating room managers/administrators help determine how to most efficiently equip their operating rooms with endoscopic equipment.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for ureteroscopy and laser lithotripsy for individual renal stones ranging in size from 5 mm to 20 mm in all intrarenal locations (If there are multiple stones present, the total stone burden in cross section should not exceed 20 mm)
* 19 years or older and able to provide informed consent

Exclusion Criteria:

* patients < 18 years
* pregnant
* patients with known nephrocalcinosis .
* any other reason that in the opinion of the investigator would make the participant unsuitable for enrollment in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Stone-free status | 6-10 weeks
  Overall kidney stone burden that remains post ureteroscopy (if any)

SECONDARY OUTCOMES:
Case completion with one scope | Day of procedure
  Was the operation able to be completed with a single scope (did the scope break and/or did another one have to be used)
Scope optics (visual quality of the image provided by the scope) | Day of procedure
  At the start and end of each procedure the surgeon will take a video clip of the intrarenal collecting system - these clips will then be evaluated and scored by blinded urologists.They will use a 5 point Likert scale that will evaluate the quality of the image in multiple categories from poor (1) to excellent (5) in multiple categories. Categories include: Focus/Sharpness, Exposure, Color Accuracy, and Overall Image Quality.
Maintenance and Repair | Through study completion, an average of 8 months
  number of cases until repair (reusable scope),
Secondary procedures and/or unanticipated clinical events | 4-6 weeks post operatively
  Includes adjuvant procedures and unscheduled hospital visits

CONTACTS AND LOCATIONS:
Overall Officials: Ben H Chew, MD, Principal Investigator — University of British Columbia, Associate Professor
Locations (2):
- Eye and Ear Institute - Department of Urology, Columbus, Ohio, United States
- University of British Columbia, Vancouver, British Columbia, Canada